CLINICAL TRIAL: NCT02184923
Title: Verticality Perception in Patients With Acute Lateralized Lesions Along the Central Graviceptive Pathways- Acute Assessment on the Ward and the Stroke Center
Brief Title: Verticality Perception in Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: verticality_percept_stroke_zrh
Record Dates: First submitted 2014-07-03; First posted 2014-07-09 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2019-12

CONDITIONS: Verticality Perception in Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- verticality measurements (Experimental)
  Interventions: Other: presentation of visual vertical

INTERVENTIONS:
Other: presentation of visual vertical

SUMMARY:
The long-term goal of this research is to advance our knowledge of how information from the labyrinth is brought to perception and how adaptation to vestibular imbalance influences spatial orientation. In healthy human subjects verticality perception is accurate while upright.The strategy of this research is to quantify changes in verticality perception after unilateral lesions along the central graviceptive pathways and to assess the frequency and pattern of abnormal verticality perception in patients with acute stroke (ischemic or hemorrhagic). Our underlying hypothesis is that screening for erroneous verticality perception by use of a mobile device assessing the subjective visual vertical (SVV) during the acute phase (i.e., within 24-48 hours after symptom onset) reliably identifies those patients with defects. Early detection of deficits in verticality perception may help to initiate balance physiotherapy early.

ELIGIBILITY:
Inclusion Criteria:

1. ages 18-90 years
2. informed consent
3. for group 1: acute (i.e. symptom onset <3 days ago) lateralized ischemia or hemorrhage as confirmed by clinical examination and / or brain imaging (CT or MRI).
4. absence of exclusion criteria

Exclusion Criteria:

1. history of a peripheral-vestibular deficit
2. disturbed consciousness
3. severe sensory or motor aphasia
4. visual field deficits
5. other neurological or systemic disorder which can cause dementia or cognitive dysfunction
6. intake of antidepressants, sedatives, or neuroleptics

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of verticality perception | during the measurement period (10 minutes)

SECONDARY OUTCOMES:
Test-re-test reliability of verticality perception | from session 1 (day 0) to session 2 (day 1)

CONTACTS AND LOCATIONS:
Overall Officials: Dominik Straumann, MD, Principal Investigator — University Hospital Zurich, Division of Neurology
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Background] Zwergal A, Rettinger N, Frenzel C, Dieterich M, Brandt T, Strupp M. A bucket of static vestibular function. Neurology. 2009 May 12;72(19):1689-92. doi: 10.1212/WNL.0b013e3181a55ecf. PMID 19433743